CLINICAL TRIAL: NCT00664976
Title: Treatment Resistant Depression in Bipolar Disorder - A Randomized Controlled Trial of Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Vest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECT-0408
Record Dates: First submitted 2008-04-14; First posted 2008-04-23 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Bipolar Disorder
Keywords: bipolar depression; Electroconvulsive therapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Electroconvulsive Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Electroconvulsive therapy
  Interventions: Procedure: Electroconvulsive therapy
- 2 (Active Comparator): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Procedure: Electroconvulsive therapy — Electroconvulsive therapy
  Arms: 1
Other: Treatment as usual — Pharmacological antidepressant as usual in the departments: Mood stabilizers as Lithium, lamotrigine, valproate, quetiapine, carbamazepine and olanzapine. Antidepressants + Psychosocial treatment as usual.
  Arms: 2

SUMMARY:
This project is a randomized controlled trial of electroconvulsive therapy (ECT) compared to treatment as usual (TAU) in the treatment of treatment resistant depression (TRD) in bipolar disorder. The purpose of the trial is to document the effect size, relative effect size and adverse effects of ECT in this condition. A specific purpose is to gain more knowledge about the effect on cognitive function.

DETAILED DESCRIPTION:
This project is a randomized controlled trial of electroconvulsive therapy (ECT) compared to treatment as usual (TAU) in the treatment of treatment resistant depression (TRD) in bipolar disorder. The purpose of the trial is to document the effect size, relative effect size and adverse effects of ECT in this condition. A specific purpose is to gain more knowledge about the effect on cognitive function.

In a national collaboration project the investigators will compare the antidepressant and cognitive effects of ECT with the effects of a drug treatment in use for this condition; a treatment algorithm combining antidepressants, mood stabilizer and antipsychotic drugs. The investigators will use a neuropsychological test battery to disclose possible ECT induced changes in cognitive function, and investigate any long-lasting changes.

In addition, several studies have implemented inflammatory processes in the pathogenesis of depression; inflammatory processes will be examined as a function of changes in clinical status and of treatment modality.

The study is a national collaboration, using the Bipolar Research And Innovation Network- BRAIN, and all the patients are included in the BRAIN-study. The study is funded by Helse Vest RHF, Regional research network on mood disorders (MoodNet) and Norwegian hospitals.

ELIGIBILITY:
Inclusion Criteria:

* ECT indicated
* Diagnosis of DSM-IV-TR of Bipolar I or Bipolar II disorder as verified by the semi-structured diagnostic interviews SCID or MINI plus.
* Severity: meet DSM-IV-TR criteria of depressive episode, MADRS of 25 or above.
* Treatment resistance
* None response to two trials (during lifetime) with mood stabilizer with proven efficacy in bipolar depression (lithium, lamotrigine, quetiapine, olanzapine) and /or antidepressants.
* A trial is defined as at least 6 weeks in adequate or tolerated dose as reported by the patient, or patients that have been unable to comply with 6 weeks trials of mood stabilizer or an antidepressant.
* Less than 50% reduction in MADRS values or still meet DSM -IV-TR criteria of depressive episode
* Inpatients the first week after start of treatment condition
* The patient are to be treated by the psychiatrist at the hospital for the whole duration of the study (6 weeks)
* Age ≥ 18
* Patient competent to give informed consent according to the judgement of the clinician
* Written informed consent
* Patient fluent in Norwegian language

Exclusion Criteria:

* Earlier ECT nonresponse
* ECT within the last six months
* More than four failed adequate medication trials in the current episode
* Rapid cycling bipolar disorder (e.g.4 or more episodes per year)
* Use of medication or substances (such as pethidine, alcohol, drugs) incompatible with drug medication or ECT. Such medication must be stopped a least 5 half-lives before inclusion in the study.
* Current use of all other psychotropic medication 5 t1/2 before inclusion and during the study period with the exception of the following:
* The use of alimemazine (max dose 30 mg daily), chlorpromazine (max dose 25 mg x 2 daily) and chlorprotixen (max dose 20 mg x 2) is allowed. The use of mianserin (max dose 10 mg daily) is allowed. Such medication has to been discontinued at least 2 days prior neuropsychological assessment. Medication related to the ECT procedure is allowed.
* Inability to comply with study protocol
* Unstable serious medical conditions, including clinically relevant laboratory abnormalities
* Conditions that affect neuropsychological assessment such as Parkinson's Disease, Multiple sclerosis, stroke, alcohol and substance abuse or dependence (according to SCID or DSM-IV-TR)
* Pregnancy or lactation
* Fertile women without adequate contraception (Adequate contraception includes: abstinence, oral contraceptives, intrauterine devices, barrier method)
* YMRS of 20 or more
* Patient at high suicidal risk according to clinicians' judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Improvement in depression | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arne Vaaler, MD PhD, Study Director — NTNU; Helse Vest RHF
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - St Olavs Hospital, Østmarka sykehus, Trondheim

REFERENCES:
- [Result] Schoeyen HK, Kessler U, Andreassen OA, Auestad BH, Bergsholm P, Malt UF, Morken G, Oedegaard KJ, Vaaler A. Treatment-resistant bipolar depression: a randomized controlled trial of electroconvulsive therapy versus algorithm-based pharmacological treatment. Am J Psychiatry. 2015 Jan;172(1):41-51. doi: 10.1176/appi.ajp.2014.13111517. Epub 2014 Oct 31. PMID 25219389
- [Derived] Bjoerke-Bertheussen J, Schoeyen H, Andreassen OA, Malt UF, Oedegaard KJ, Morken G, Sundet K, Vaaler AE, Auestad B, Kessler U. Right unilateral electroconvulsive therapy does not cause more cognitive impairment than pharmacologic treatment in treatment-resistant bipolar depression: A 6-month randomized controlled trial follow-up study. Bipolar Disord. 2018 Sep;20(6):531-538. doi: 10.1111/bdi.12594. Epub 2017 Dec 21. PMID 29267990
- [Derived] Kessler U, Schoeyen HK, Andreassen OA, Eide GE, Malt UF, Oedegaard KJ, Morken G, Sundet K, Vaaler AE. The effect of electroconvulsive therapy on neurocognitive function in treatment-resistant bipolar disorder depression. J Clin Psychiatry. 2014 Nov;75(11):e1306-13. doi: 10.4088/JCP.13m08960. PMID 25470096
- [Derived] Kessler U, Schoeyen HK, Andreassen OA, Eide GE, Hammar A, Malt UF, Oedegaard KJ, Morken G, Sundet K, Vaaler AE. Neurocognitive profiles in treatment-resistant bipolar I and bipolar II disorder depression. BMC Psychiatry. 2013 Apr 4;13:105. doi: 10.1186/1471-244X-13-105. PMID 23557429
- [Derived] Kessler U, Vaaler AE, Schoyen H, Oedegaard KJ, Bergsholm P, Andreassen OA, Malt UF, Morken G. The study protocol of the Norwegian randomized controlled trial of electroconvulsive therapy in treatment resistant depression in bipolar disorder. BMC Psychiatry. 2010 Feb 23;10:16. doi: 10.1186/1471-244X-10-16. PMID 20178636